CLINICAL TRIAL: NCT03298412
Title: A Phase 2 Open-Label Study to Determine the Effect of Blinatumomab on Minimal Residual Disease in Subjects With High-risk Diffuse Large B-cell Lymphoma Post-autologous Hematopoietic Stem-cell Transplantation.
Brief Title: Effect of Blinatumomab on Minimal Residual Disease (MRD) in Diffuse Large B-Cell Lymphoma (DLBCL) Subjects Post Autologous Hematopoietic Stem Cell Transplantation (aHSCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early Closure due to rare patient population
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150291; 2016-003255-30 (EudraCT Number)
Record Dates: First submitted 2017-09-12; First posted 2017-10-02 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: High-risk Diffuse Large B-cell Lymphoma
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): After a run-in period of up to 24 months to evaluate MRD status and assess eligibility for treatment assignment, participants received blinatumomab intravenous (IV) infusion at an initial dose of 9 μg/day for the first 7 days of treatment, escalated (dose-step) to 28 μg/day starting on Day 8 (Week 2), followed by a dose-step to 112 μg/day starting on Day 15 (Week 3) and continuing until completion of therapy (Day 57 of Cycle 1).
  Cycle 1 of blinatumomab treatment is 12 weeks (84 days) in duration and includes 8 weeks (56 days) of blinatumomab IV infusion followed by a 4-week (28-day) treatment-free interval.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab is administered as a continuous IV infusion.
  Other Names: BLINCYTO; AMG 103

SUMMARY:
The study will estimate the MRD-negative response rate after treatment with blinatumomab in subjects with high-risk DLBCL who are MRD-positive following aHSCT. The clinical hypothesis is that the MRD-negative response rate will be greater than 10%. Achieving an MRD-negative response rate of 30% would be of scientific and clinical interest.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label, single arm estimation study in adult subjects with high-risk DLBCL in complete remission. The study will consist of up to a 28-day screening period, a run-in period of up to 24 months, a 12-week treatment period (8 weeks of blinatumomab treatment followed by a 4-week treatment free period), a 30-day safety follow-up visit after the last dose of blinatumomab, and a long-term follow-up period that begins after the safety follow-up visit is completed until 1 year from the first dose of blinatumomab. The study will enroll approximately 90 subjects in the screening period with biopsy proven, high-risk DLBCL that are positron emission tomography-computer tomography (PET-CT) negative 90 days (± 30 days) post aHSCT. During the run-in period subjects will be followed by clinic visits at regular interval for up to 24 months for monitoring of MRD status in plasma by a next generation sequencing (NGS)-based assay. It is estimated 30 subjects will be either MRD-positive at screening or become MRD-positive during the 24-month run-in period. The number of subjects enrolled may be altered in order to ensure that approximately 30 subjects are assigned to treatment with blinatumomab. Enrollment may be stopped, once approximately 30 subjects have been assigned to treatment with blinatumomab.

ELIGIBILITY:
Inclusion and Exclusion Criteria - Part 1

Inclusion Criteria - Part 1

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures or subject's legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
* Age ≥ 18 at time of informed consent
* Biopsy-proven DLBCL excluding DLBCL that represents transformation of indolent non-Hodgkin's lymphoma (NHL) Note: Lymphoblastic Lymphoma and Burkitt Lymphoma histology are not eligible
* Subject has ≥ 1 characteristic feature of high-risk DLBCL:

  * High-risk first complete remission (defined as interim positron emission tomography - computed tomography (PET-CT) positive or < complete remission to frontline chemotherapy AND achieved complete remission to platinum-containing salvage)
  * Relapse within 1 year of diagnosis
  * Secondary age-adjusted international prognostic index > 1
  * Partial response/partial metabolic response after minimum of 2 cycles of platinum-containing salvage chemotherapy
  * C-myc rearrangement
* aHSCT with high-dose chemotherapy following first (or later) salvage treatment.
* PET-CT negative (Deauville score ≤ 3) 90 days (± 30 days) post aHSCT
* Available relapsed and/or diagnostic pathology formalin-fixed paraffin-embedded (FFPE) tumor block or slide samples at the time of enrollment including the successful identification of malignant clone sequences by the central laboratory.
* MRD plasma sample collected ≤ 3 weeks after the post aHSCT PET-CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate organ function determined ≤ 3 weeks prior to enrollment defined as follows:

  * Hematological:

Absolute neutrophil count (ANC) ≥ 1.0 x 109/L Platelet count ≥ 75 x 109/L Hemoglobin ≥ 8 g/dL

* Renal:

Creatinine clearance ≥ 50 mL/min Cockcroft-Gault equation

* Hepatic:

Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN) Total bilirubin < 2 x ULN (unless Gilbert's Disease or if liver involvement with lymphoma)

* Subject will be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge including but not limited to:
* Completion of up to a 24-month run-in period
* Completion of all regularly scheduled study visits including blood draws for MRD assessment, clinical disease state assessment, PET-CT scans (ie, at time of MRD positivity or relapse), assignment to treatment with blinatumomab

  * Other Inclusion criteria may apply. See "Inclusion and Exclusion criteria - Part 2".

Exclusion Criteria - Part 1

* Clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia,stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, and psychosis
* Evidence of CNS involvement with DLBCL at disease evaluation obtained prior to starting blinatumomab
* Current autoimmune disease or history of autoimmune disease with potential of CNS involvement
* Prior anti-CD19 directed therapies
* Prior alloHSCT
* Received radiation ≤ 2 weeks prior to enrollment
* Infection with human immunodeficiency virus or chronic infection with hepatitis B virus (hepatitis B surface antigen positive) or hepatitis C virus (anti-hepatitis C virus positive)
* History of malignancy other than DLBCL within the past 3 years with the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
* Subject has known hypersensitivity to immunoglobulins or any of the products or components to be administered during dosing.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Women who are pregnant or breastfeeding or planning to become pregnant or breastfeed while receiving blinatumomab and for an additional 48 hours after the last treatment dose of blinatumomab. (Females of child bearing potential should only be included after a negative highly sensitive urine or serum pregnancy test.)
* Women of childbearing potential unwilling to use an acceptable method of effective contraception while receiving blinatumomab and for an additional 48 hours after last dose of blinatumomab. Note: The pregnancy, breastfeeding and contraceptive requirements are specific to blinatumomab. The investigator is responsible for providing the subject (male and female) with pregnancy and breastfeeding (female only) avoidance requirements for other medications given during the study.
* Currently receiving treatment in another investigational device or drug study or less than 30 days since ending treatment on another investigational device or drug study. Other investigational procedures while participating in this study are excluded.

  * Other Exclusion criteria may apply. See "Inclusion and Exclusion criteria - Part 2".

Inclusion and Exclusion Criteria - Part 2

Inclusion Criteria - Part 2

* MRD-positive assessment (by NGS analysis) at enrollment or at any time during the run-in 1 period
* PET-CT negative (defined by Deauville criteria ≤ 3) at run-in 2 performed ≤ 3 weeks from MRD test result available to the site at run-in 1. Historical PET-CT are allowed if performed ≤ 6 weeks from day 1 (first dose of blinatumomab) and subject has no clinical signs or symptoms suggestive of disease progression (eg, increase in lactate dehydrogenase [LDH] not otherwise explained)
* Adequate organ function determined ≤ 7 days prior to treatment assignment with blinatumomab as follows:

  * Hematological:

ANC ≥ 1.0 x 109/L Hemoglobin ≥ 8 g/L Platelet count ≥ 75 x 109/L

* Renal:

Creatinine clearance ≥ 50 mL/min Cockcroft-Gault equation

* Hepatic:

AST and ALT < 3 x ULN Total bilirubin < 2 x ULN (unless Gilbert's Disease or if liver involvement with lymphoma)

Exclusion Criteria - Part 2

* Subject has active infection requiring systemic therapy
* Any change in the part 1 eligibility criteria during the run-in period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- United States (4):
  - Research Site, Atlanta, Georgia
  - Research Site, Maywood, Illinois
  - Research Site, Cleveland, Ohio
  - Research Site, Dallas, Texas
- Australia (4):
  - Research Site, St Leonards, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Clayton, Victoria
  - Research Site, Geelong, Victoria
- Belgium (3):
  - Research Site, Charleroi
  - Research Site, Leuven
  - Research Site, Liège
- France (8):
  - Research Site, Créteil
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Rouen
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Italy (6):
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Torino
- Switzerland (4):
  - Research Site, Bellinzona
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants from Australia, France, Greece, Italy, Switzerland, and the United States. The first participant enrolled on 23 May 2018, and the last participant enrolled on 05 August 2019.
Pre-assignment Details: The study included a Screening period (up to 28 days), and a run-in period of up to 24 months to evaluate minimal residual disease (MRD) status and assess eligibility for treatment assignment.
Period: Run-in Period
Arm/Group | Blinatumomab
Started | 10
Completed | 1
Not Completed | 9
Not completed — Other, Not Specified | 1
Not completed — Disease Progression | 1
Not completed — Ineligibility Determined | 1
Not completed — Decision by Sponsor | 6
Period: Treatment Period
Arm/Group | Blinatumomab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: MRD-Negative Rate at the End of Cycle 1
Description: The estimated MRD-negative rate, calculated as the percentage of participants with MRD-negative status after treatment with blinatumomab. MRD-negative status was assessed by positron emission tomography-computed tomography (PET-CT) or computed tomography (CT).
Time Frame: 12 weeks (84 days)
Population: Full analysis set (all participants who received any infusion of blinatumomab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 1
percentage of participants | 100 [2.5 to 100]

2. Secondary Outcome: Kaplan-Meier Estimate: Progression-Free Survival (PFS)
Description: PFS, calculated as the time from the date of first dose of blinatumomab until the date of diagnosis of relapse of lymphoma (by PET-CT, CT, clinical assessment or relapse biopsy, whichever was the preferred method), or date of death, whichever was earliest. Participants who were alive and who did not have progression or new anti-tumor treatment (excluding any stem cell transplantation) were to be censored at last date of tumor assessment.
Time Frame: up to 1 year from first dose of blinatumomab
Population: Full analysis set (all participants who received any infusion of blinatumomab).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 1
months | NA [NA to NA] — NA=Not estimable (1 participant in analysis set).

3. Secondary Outcome: Kaplan-Meier Estimate: Duration of MRD-Negative Status
Description: The duration of MRD-negative status, assessed only in participants who achieve MRD-negative status after blinatumomab treatment, was defined as the time when a negative MRD result was first established until documented MRD-positive re-occurrence, disease progression or, death due to any cause. Participants without any of these events at the time of the analysis were to be censored at their last disease assessment date. MRD-negative status was assessed by PET-CT or CT.
Time Frame: up to 1 year from first dose of blinatumomab
Population: Full analysis set (all participants who received any infusion of blinatumomab).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 1
months | 10.26 [NA to NA] — NA=Not estimable (1 participant in analysis set).

4. Secondary Outcome: Kaplan-Meier Estimate: Overall Survival (OS)
Description: OS, defined as time from the first dose of blinatumomab treatment until death due to any cause. Participants still alive at the time of the analysis were censored at date last known to be alive.
Time Frame: up to 1 year from first dose of blinatumomab
Population: Full analysis set (all participants who received any infusion of blinatumomab).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 1
months | NA [NA to NA] — NA=Not estimable (1 participant in analysis set).

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence. A serious AE is defined as an AE that is: fatal; life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; a congenital anomaly/birth defect; other medically important serious event. TEAEs are events with an onset after the administration of the first dose of blinatumomab treatment through 30 days after the end of blinatumomab treatment. Events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE): Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), Grade 5 (death).
Time Frame: From first dose of study drug through 30 days after the last dose of study drug. The treatment duration for the participant who received blinatumomab was 57 days.
Population: Full Analysis Set: all participants who received at least 1 dose of blinatumomab.
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 1
participants
  Any TEAE | 1
  Grade 3 TEAE | 1
  Serious TEAE | 0
  TEAE Leading to Study Drug Discontinuation | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrollment through 24 months of run-in period among participants who did not receive study drug, or through 1 year after the first dose of study drug, or end of study. SAEs/AEs were collected from first dose of study drug through 30 days after the last dose of study drug. The treatment duration for the participant who received blinatumomab was 57 days.
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=1)
Neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03298412/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT03298412/SAP_001.pdf